CLINICAL TRIAL: NCT06478680
Title: Comparing Effects of Conventional Neurorehabilitation With Exoskeleton With High-intensity Gait Training on Gait, Balance, and Depression Following Stroke and the Impact of Social Determinants of Health and Depression on Patients' Adherence to Physical Therapy
Brief Title: Comparing Effects of Conventional Neurorehabilitation With Exoskeleton With High-intensity Gait Training
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participants
Sponsor: Alvernia University (Other)
Collaborators: Good Shepherd Rehabilitation Network (Other)
Responsible Party: Principal Investigator, Soo Yeon Sun, PT, PhD, Associate professor, Alvernia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2176775-1
Record Dates: First submitted 2024-06-23; First posted 2024-06-27 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Gait, Hemiplegic
Keywords: health literacy; balance; compliance to therapy; gait function; high intensity gait training; exoskeleton
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High intensity gait training (Active Comparator): One session of conventional neurorehabilitation intervention per week One session of Forward Walking with EksoGT per week
  Interventions: Behavioral: High intensity gait training
- Exoskeleton mediated gait training (Experimental): Two sessions of High-Intensity Gait Training
  Interventions: Behavioral: Exoskeleton mediated gait training

INTERVENTIONS:
Behavioral: Exoskeleton mediated gait training — 1 session of Forward Walking with EksoGT per week
  1 session of conventional neurorehabilitation intervention per week
  * Transfer training
  * Gait training
  * Balance (sitting/standing; static/dynamic)
  * Strength
  * Neuromuscular re-education
  * Orthotics
  * Positioning
  * Caregiver education
  * Assistive device
  * Wheelchair assessment and mobility
  * Endurance training
  Other Names: EksoGT-mediated gait training
  Arms: Exoskeleton mediated gait training
Behavioral: High intensity gait training — 2 sessions of High-Intensity Gait Training at a target heart rate of 60-80% of the maximum heart rate or target RPE of 15-18
  * Forward stepping practice
  * Backwards stepping practices
  * Sidestepping
  * Stairs
  * Balance and compliant surface training while walking
  * Propulsion
  * Lateral balance training
  * Stability training
  * Stance control training
  * Limb advancement
  Arms: High intensity gait training

SUMMARY:
The purpose of this research is to compare improvements between the rehab intervention with walking practice using the robotic exoskeleton versus walking practice that is vigorous enough to keep participants' heart rate over a certain target level during physical therapy sessions. Investigators want to compare improvements in your walking function and mental health that occur after 20 interventions. The study also aims to evaluate if participants' mental health, social support, and health literacy affect attendance at physical therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English or Spanish-speaking
* A diagnosis of stroke (intracerebral hemorrhage or acute ischemic stroke)
* Referred to Good Shepherd Rehabilitation Outpatient Physical Therapy Clinic

Exclusion Criteria:

* Unable to follow 1-step commands
* > 220 pounds (100 kg)
* Height < 5'0" or > 6'4"
* Unable to take a few steps with assistance
* A score of ≥ 50/56 on Berg Balance Scale (BBS)
* A score of ≥ 26/30 on Functional Gait Assessment (FGA)
* Resting blood pressure >180/110 mmHg
* Resting heart rate > 120 bpm
* Severe cardiac disease (New York Heart Association Classification IV)
* Severe spasticity (Modified Ashworth score > 3)
* Unstable spine or unhealed pelvic/limb fractures
* Active heterotrophic ossification impacting lower extremity range of motion
* Significant lower or upper extremity contractures
* Inability to achieve neutral ankle dorsiflexion with 12° of knee flexion
* Pregnancy
* Colostomy
* Poor skin integrity in areas in contact with the EksoGTTM
* Unresolved deep vein thrombosis
* Lower limb prosthesis or amputation
* Leg length discrepancies > 0.5 inches for upper legs, 0.75 inches for lower legs
* ROM restrictions preventing normal, reciprocal gait
* Inability to stand for > 3 minutes due to pain or orthostatic hypotension
* Pusher syndrome
* Cortical blindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Demographic Questionnaire | Pre-intervention
  Questions include age, sex, date of birth, race/ethnicity, total income during T the past 12 months, main occupation and when was the last work, language at home, marital status, education level, and if they take any antidepressants.
Newest Vital Sign (NVS) | Pre-intervention
  The NVS is a 6-question screening tool that identifies participants' risk of low or limited health literacy (HL) based on interpreting an ice cream nutrition label.
Multidimensional Scale of Perceived Social Support (MSPSS) | Pre-intervention
  The Multidimensional Scale of Perceived Social Support is a 12-item self-administered scale that measures social support. The total score for the MSPSS ranges from 12 to 84, with higher scores indicating higher levels of perceived social support.
Patient Health Questionnaire (PHQ-9) | Pre-intervention, After 10 interventions (~5 weeks), After 20 interventions (~10 weeks)
  The PHQ-9 is a self-administered depression screening tool with nine items. It has been reported that the PHQ-9 is the best-performing tool for screening for post-stroke depression.
3-Meter Backwards Walk Test (3MBWT) | Pre-intervention, After 10 interventions (~5 weeks), After 20 interventions (~10 weeks)
  The 3MBWT measures the time (in seconds) it takes for a participant to walk 3 meters backward, hence assessing a backward gait speed. Backward gait speed is used to evaluate neuromuscular control, proprioception, protective reflexes, fall risk, and balance. Use of assistive devices will be documented.
6-Minute Walk Test | Pre-intervention, After 10 interventions (~5 weeks), After 20 interventions (~10 weeks)
  The 6MWT assesses participants' aerobic capacity/endurance by recording the distance (in meters) that the participants walk in 6 minutes. Assistive devices may be used and will be documented.
10-meter Walk Test | Pre-intervention, After 10 interventions (~5 weeks), After 20 interventions (~10 weeks)
  The 10mWT assesses walking speed in meters/second (m/s) over a short distance (10m). Two trials are administered at the patient's comfortable walking speed, followed by 2 trials at their fast walking speed, per Physical Therapist's instruction. The 2 trials for each speed are then averaged and the 2 gait speeds (preferred and fast) are documented in m/s. Assistive devices may be used, and will be documented.
Muscle coactivation index | Pre-intervention, After 10 interventions (~5 weeks), After 20 interventions (~10 weeks)
  Muscle coactivation index will be calculated based on the EMG signals from 8 leg muscles (bilateral tibialis anterior, medial gastrocnemius, rectus femoris, medial hamstring). Surface electromyographic recordings will be conducted during forward and backward walking tests.
Berg Balance Scale (BBS) | Pre-intervention, After 10 interventions (~5 weeks), After 20 interventions (~10 weeks)
  The Berg Balance Scale is a 14-item clinician-rated measure that assesses static and balance in sitting and standing. It has a maximum score of 56 points. Each item is scored on a 5-point scale from 0 to 4, with 0 indicating the subject is unable to perform the task and 4 being the highest score.
Functional Gait Assessment (FGA) | Pre-intervention, After 10 interventions (~5 weeks), After 20 interventions (~10 weeks)
  The FGA is used to assess postural stability during walking and assesses an individual's ability to perform multiple motor tasks while walking. The Functional Gait Assessment (FGA) is scored on a 4-point ordinal scale ranging from 0-3, with 0 indicating severe impairment and 3 indicating normal ambulation. The total score is calculated by summing all the items and ranges from 0-30, with lower scores indicating greater impairment.
Borg rating scale of Perceived Exertion | Pre-intervention, After 10 interventions (~5 weeks), After 20 interventions (~10 weeks)
  The Borg Rating Scale of Perceived Exertion will be measured in all participants at the completion of 6 minute walk test. It measures exertion on a scale of 0 (no exertion or resting) to 10 (pushing oneself to the max).

SECONDARY OUTCOMES:
Patient compliance | After 20 interventions (~10 weeks)
  Patient attendance to physical therapy is tracked and will be measured as >80% attendance to physical therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Yeon Sun, PhD, Principal Investigator — Alvernia University; Kelley Limbauan, PT, DPT, NCS, Principal Investigator — Good Shepherd Rehabilitation Network
Locations (1):
- Good Shepherd Rehabilitation, Allentown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No